CLINICAL TRIAL: NCT05754541
Title: Guo's Endovascular Aortic Arch Replacement of Aortic Dissection by WeFlow-Tribranch Endoprothesis: a Multicenter Pilot Study(Graft Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WeFlow-Tribranch V1.0
Record Dates: First submitted 2023-02-07; First posted 2023-03-06 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-07

CONDITIONS: Aortic Aneurysm and Dissection
Keywords: Stent Graft
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WeFlow-Tribranch Aortic Arch Stent Graft System (Experimental)
  Interventions: Device: WeFlow-Tribranch Aortic Arch Stent Graft System

INTERVENTIONS:
Device: WeFlow-Tribranch Aortic Arch Stent Graft System — Endovascular treament in patients with aortic arch dissection and aneurysm by WeFlow-Tribranch Aortic Arch Stent Graft System

SUMMARY:
To explore the effect and prognosis of endovascular interventional therapy in high-risk patients with aortic arch dissection and aneurysm

DETAILED DESCRIPTION:
The WeFlow-Tribranch Aortic Arch Stent Graft System first in man study is a prospective, multi-center, single arm trial, which will enroll a total of 20 patients. The goal of this study is to evaluate the safety and efficacy of WeFlow-Tribranch Aortic Arch Stent Graft System in the treatment of patients with aortic arch dissection and aneurysm.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years old.
2. The patient was diagnosed with subacute or chronic aortic arch dissection, or Aortic arch aneurysms.
3. Patients showing a suitable vascular condition, including:

   1. Ascending aorta length greater than 50 mm (from the aortic sinusoid junction to the proximal cardiac margin of the innominate artery).
   2. Ascending aorta diameter ≥ 24 mm and ≤ 48 mm;
   3. Proximal anchoring zone length ≥ 30 mm;
   4. Innominate artery diameter ≤ 24 mm and ≥ 7 mm, length ≥ 20 mm；
   5. Left common carotid artery or left subclavian artery diameter ≤ 24 mm and ≥ 7 mm, length ≥ 20 mm；
   6. Suitable arterial access for endovascular interventional treatment ;
4. Patients able to understand the purpose of the trial, participate in the trial voluntarily with informed consent form signed by the subject him/herself or his or her legal representative, and willing to complete follow-up visits as required under the protocol.
5. Patients evaluated by at least two vascular surgeons or cardiac surgeons as high surgical risk patients or deemed to have significant surgical contraindications. (The recommended reference criteria are: EuroSCORE score ≥ 6, or CFS score > 4, or ASA grade 3-4, or there are other high-risk surgical factors that affect the prognosis of the subject, such as patients with a history of open surgery, other high-risk factors judged by a physician team, or patients who refuse open surgery.)

Exclusion Criteria:

1. Patients that have experienced systemic infection during past three months;
2. Neck surgery was performed within three months;
3. Infectious aortic disease、Takayasu arteritis，Marfan syndrome (or other connective tissue diseases );
4. Patients with severe stenosis, calcification, thrombosis or tortuosity of the Brachiocephalic trunk, Left common carotid artery or left subclavian artery;
5. Heart transplant patients;
6. Patients that have suffered MI or stroke during past three months;
7. Patients with Class IV heart function (NYHA classification) or LVEF<30%
8. Active peptic ulcers or upper gastrointestinal bleeding occurring within the previous three months;
9. Hematological abnormality, defined as follows: Leukopenia (WBC < 3 × 109/L), acute anemia (Hb < 90 g/L); thrombocytopenia (PLT count < 50 × 109/L);
10. Patients with renal insufficiency， serum creatinine > 150 umol/l (or 3.0 mg/dl) and / or end-stage renal disease requiring renal dialysis shall be determined by the investigator after comprehensive analysis;
11. Subjects with severe liver dysfunction and ALT or AST exceeding 3 times the upper limit of normal; Subjects whose serum total bilirubin (STB) exceeds 2 times the upper limit of normal;
12. Patients with intestinal necrosis and lower limb ischemic necrosis;
13. Paraplegic patients;
14. Patients that are pregnant or breastfeeding;
15. Patients with allergies to contrast agents;
16. Patients with a life expectancy of less than 12 months;
17. Patients currently participating in other drug or device research;
18. Any other disease or abnormality that the investigators believe may hinder endovascular interventional treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality and major stroke within 12 months after surgery. | 12 months post-intervention
  All-cause mortality includes cardiac mortality, non-cardiac mortality and mortality from unknown causes. Severe stroke is defined as a modified Rankin score (mRS) ≥ 2 at 90 days following stroke onset

SECONDARY OUTCOMES:
Aortic-related mortality within 12 months post operation. | within 12 months post operation
  Refers to mortality caused by a ruptured aortic dissection/aneurysm or endovascular interventional treatment.
Aortic remodeling results. | 1 month, 6 months and 12 months post-intervention
  Compare the results of CTA before operation and on the 30th day, 6th month and 12th month after operation, the expansion of the true lumen and the thrombosis of the false lumen at the coverage of the aortic dissection vascular stent to determine whether the blood vessel is successfully remodeled，or CTA reexamination 12 months after operation showed that the maximum diameter of Aortic aneurysm increased by ≤ 5 mm compared with that before operation.
Major adverse events occurring within 30 days after surgery. | within 30 days after surgery
  Refers to all-cause mortality, myocardial infarction, ischemic stroke or respiratory failure occurring within 30 days after surgery. More specifically, myocardial infarction refers to a drastic reduction or complete interruption of the coronary blood supply due to coronary artery disease, resulting in severe and prolonged acute ischemia of the corresponding myocardium, leading to necrosis of cardiomyocytes. Ischemic stroke refers to the end result of necrosis of brain tissue caused by narrowing or occlusion of the arteries supplying blood to the brain or insufficient blood supply to the brain. Respiratory failure is defined as a state resulting in significantly prolonged intubation, tracheotomy, deterioration of lung function, or other fatal outcomes.
Incidence of severe adverse events. | within 12 months post-intervention
  Refers to an event that occurs during the clinical trial that results in mortality or serious deterioration in patient health, including a fatal illness or injury, a permanent defect in body structure or body function, or an event that requires medical or surgical intervention to avoid one or more permanent defects in body structure or body function.

CONTACTS AND LOCATIONS:
Overall Officials: wei Guo, Principal Investigator — Chinese PLA Gencral Hosptial
Locations (4):
- China (4):
  - Chinese PLA Gencral Hosptial, Beijing, Beijing Municipality
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No